CLINICAL TRIAL: NCT01455831
Title: A Multicentre Randomized Controlled Trial of the Use of Extended Peri-Operative Low Molecular Weight Heparin to Improve Cancer Specific Survival Following Surgical Resection of Colorectal Cancer
Brief Title: Extended Peri-operative Tinzaparin to Improve Disease-free Survival in Patients With Resectable Colorectal Cancer
Acronym: PERIOP-01
Status: Completed | Phase: Phase 3 | Type: Interventional
Sponsor: Ottawa Hospital Research Institute (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Prevention
Other Study IDs: 221097
Record Dates: First submitted 2011-10-18; First posted 2011-10-20 (Estimated); Last update posted 2021-05-17 (Actual); Status verified 2021-05

CONDITIONS: Adenocarcinoma of the Colon
MeSH Terms: conditions — Colonic Neoplasms | interventions — Tinzaparin

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- Extended peri-operative thromboprophylaxis (Experimental): The experimental arm will receive a subcutaneous injection of 4,500 IU of tinzaparin daily beginning at randomization and continued for 56 days following resection. There will be a minimum of one dose of pre-operative LMWH since it is not reasonable to delay surgery for the purpose of administering LMWH. The maximum duration of pre-operative LMWH will be 6 weeks.
  Interventions: Drug: Tinzaparin
- Standard thromboprophylaxis (Active Comparator): The control arm will receive a daily subcutaneous injection of 4,500 IU of tinzaparin beginning with the first post-operative dose and continued for the duration of hospitalization.
  Interventions: Drug: Tinzaparin

INTERVENTIONS:
Drug: Tinzaparin — The experimental arm will receive a subcutaneous injection of 4,500 IU of tinzaparin daily beginning at randomization and continued for 56 days following resection. There will be a minimum of one dose of pre-operative LMWH since it is not reasonable to delay surgery for the purpose of administering LMWH. The maximum duration of pre-operative LMWH will be 6 weeks.
  Other Names: Innohep
  Arms: Extended peri-operative thromboprophylaxis
Drug: Tinzaparin — The control arm will receive a daily subcutaneous injection of 4,500 IU of tinzaparin beginning with the first post-operative dose and continued for the duration of hospitalization.
  Other Names: Innohep
  Arms: Standard thromboprophylaxis

SUMMARY:
The human body has a natural stress response to surgery, including the formation of blood clots. This response to surgery has been shown to increase metastases (the spread of cancer cells to other organs in the body). These metastases cannot be seen at the time of surgery but when they grow into new tumors, the cancer has recurred (come back). A blood thinner called "low molecular weight heparin" (LMWH) can suppress the development of metastases after surgery in animal experiments. The investigators want to see if giving patients with colorectal cancer the blood thinner, LMWH, around the time of surgery can decrease the chance of their cancer spreading to other organs (metastases) and coming back (recurrence).

The investigators need 1075 patients to answer our scientific question. Patients who give informed consent will be randomly put into one of two groups, the experimental group and the control group. The patients in the control group will be treated with LMWH starting a few hours after surgery and every day until they leave the hospital. This is how most patients are treated after colon cancer surgery (standard care). The patients in the experimental group will be treated with LMWH for a longer period of time, starting on the day they agree to have surgery and continuing for two months after surgery. All the patients will be followed for at least three years after surgery to find out if their cancer has recurred (come back). If LMWH treatment around the time of surgery reduces the chance of recurrence in patients with colorectal cancer, it would improve the health and quality of life for these patients.

ELIGIBILITY:
Inclusion Criteria:

1. Diagnosis of pathologically-confirmed invasive adenocarcinoma of the colon or rectum
2. Pre-operative work-up that reveals potential resectability (CT scan or MRI of the abdomen and pelvis) with resection planned within 6 weeks of date of randomization
3. Pre-operative work-up that reveals no evidence of metastatic disease (CT scan or MRI of the abdomen and pelvis and chest X-ray (CXR) or CT scan of the chest)
4. Age ≥18 years
5. Hemoglobin ≥ 80g/L
6. Able and willing to comply with study procedures and follow-up examinations contained within the written consent form.

Exclusion Criteria:

1. Carcinoma only present in a completely excised polyp (i.e. no residual tumour evident in the colon)
2. Prior VTE including deep vein thrombosis (DVT) or pulmonary embolism (PE)
3. Requirement for full dose peri-operative anticoagulation
4. Contraindication to heparin therapy

   1. history of heparin induced thrombocytopenia (HIT)
   2. platelet count of less than 100 x 109/L
   3. actively bleeding
   4. severe hypertension (SBP >200 and/or DBP >120) on more than one reading
   5. documented peptic ulcer within 6 weeks
   6. severe hepatic failure (INR >1.8)
   7. creatinine clearance of < 30 ml/min as calculated by the Cockcroft-Gault formula
   8. Other contraindication to anticoagulation
5. Participating in another interventional trial that may result in co-intervention or contamination (to be determined by sponsor)
6. History of other malignancies (except for adequately treated basal or squamous cell carcinoma or carcinoma in situ) within 5 years of the colorectal cancer diagnosis
7. Pregnant or lactating
8. Unable/unwilling to providing informed consent.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 616 (Actual)
Dates: Start 2011-09; Primary Completion 2020-12-31 (Actual); Study Completion 2021-02-01 (Actual)

PRIMARY OUTCOMES:
Disease Free Survival | measured at 3 years
  Disease free survival is measured from the time of randomization until local disease recurrence, distant disease recurrence, a new primary colon cancer malignancy, other second primary cancer or death from any cause.

SECONDARY OUTCOMES:
Overall Survival | measured at 5 years
  Death from any cause
Venous Thromboembolism events | From randomization until 56 days post-surgery
  • VTE events defined as:
  a. Deep vein thrombosis: i. non-compressibility of any vein segment from the common femoral vein to the trifurcation of the popliteal vein on compressive ultrasonography ii.persistent intra-luminal filling defect of the iliac, common femoral, superficial femoral, popliteal, posterior tibial or peroneal veins on contrast venography b. Pulmonary embolism: i.high probability V/Q scan ii.positive pulmonary angiogram iii.spiral CT demonstrating intraluminal filling defect in a vessel larger than a segmental artery
Major surgical site bleeding events | From randomization until 56 days post-surgery
  • Major surgical site bleeding events defined as bleeding at the surgical site associated with:
  1. requirement for ≥4 units of packed red blood cells
  2. a drop in Hb of >40 g/L during the first post-op week
  3. bleeding requiring re-operation
  4. fatal bleeding
Major bleeding events (not including the surgical site) | From randomization until 56 days post-surgery
  • Major bleeding events (not including the surgical site) defined as:
  1. fatal bleeding, and/or
  2. symptomatic bleeding in a critical area or organ, such as intracranial, intraspinal, intraocular, retroperitoneal, intraarticular or pericardial, or intramuscular with compartment syndrome, and/or,
  3. bleeding causing a fall in hemoglobin level of ≥20 g/L, or leading to transfusion of ≥2 units of whole blood or red cells.
• Clinically relevant bleeding events prior to surgery and during the • Clinically relevant bleeding events | From randomization to 56 days post-surgery
  Clinically relevant bleeding events prior to surgery and during the follow-up period will be defined as overt bleeding episodes not meeting the inclusion for major bleeding but associated with one of the following:
  1. medical intervention;
  2. an unscheduled contact with a physician;
  3. temporary cessation of anticoagulant treatment
Transfusion requirements | From randomization to 56 days post-surgery
  Transfusion requirements using the number of units transfused:
  1. Red blood cells
  2. Platelets (Adult dose)
  3. Frozen Plasma
Correlative endpoints | 5 years
  The correlative endpoints seek to evaluate the pro-metastatic mechanisms of surgery and the antimetastatic mechanisms of LMWH in subjects undergoing surgical resection for colon cancer.
Other post-operative (day 0 - day 28) complications | Measured from Day 0 until day 28 post-operatively
  Other post-operative (day 0 - day 28) complications as defined using the modified Clavien Classification

CONTACTS AND LOCATIONS:
Overall Officials: Marc Carrier, MD, Principal Investigator — Ottawa Hospital Research Institute; Rebecca Ann Auer, MD, Principal Investigator — Ottawa Hospital Research Institute
Locations (16):
- Ghent University Hospital, Ghent, Belgium
- Canada (14):
  - Health Sciences North, Greater Sudbury, Ontario
  - Hamilton Health Sciences Corporation, Hamilton, Ontario
  - Kingston General Hospital, Kingston, Ontario
  - London Health Research Institute, London, Ontario
  - The Ottawa Hospital, Ottawa, Ontario
  - Montfort Hospital, Ottawa, Ontario
  - Queensway Carleton Hospital, Ottawa, Ontario
  - Sault Area Hospital, Sault Ste. Marie, Ontario
  - Humber River Hospital, Toronto, Ontario
  - Mount Sinai Hospital, Toronto, Ontario
  - North York General Hospital, Toronto, Ontario
  - St. Joseph's Health Centre, Toronto, Ontario
  - Sunnybrook Health Science Centre, Toronto, Ontario
  - Jewish General Hospital, Montreal, Quebec
- CHRU Brest, Brest, France

REFERENCES:
- [Derived] Auer RC, Ott M, Karanicolas P, Brackstone MR, Ashamalla S, Weaver J, Tagalakis V, Boutros M, Stotland P, Marulanda AC, Moloo H, Jayaraman S, Patel S, Le Gal G, Spadafora S, MacLellan S, Trottier D, Jonker D, Asmis T, Mallick R, Pecarskie A, Ramsay T, Carrier M; PERIOP-01 investigators. Efficacy and safety of extended duration to perioperative thromboprophylaxis with low molecular weight heparin on disease-free survival after surgical resection of colorectal cancer (PERIOP-01): multicentre, open label, randomised controlled trial. BMJ. 2022 Sep 13;378:e071375. doi: 10.1136/bmj-2022-071375. PMID 36100263